CLINICAL TRIAL: NCT04367896
Title: COVID-19 OUTBREAK AND SOLID ORGAN TRANSPLANTATION (SOT) : AN INTERNATIONAL WEB-BASED SURVEY
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: Covid-19_V1
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: COVID-19 OUTBREAK AND SOLID ORGAN TRANSPLANTATION
Keywords: COVID-19; Solid Organ Transplantation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey Group — The survey sought to elucidate equity principles that are influencing transplant decision making. The group of respondents included solid organ transplant doctors (surgeons, referring doctors, transplant physicians, transplant coordinators, ICU transplant doctors), COVID-doctors (ICU doctors, Infectious Disease Doctors, Pulmonologists, Internists), and Ethicists with experience of transplant related issues.
  Respondent identification:
  A. The e-mail addresses of corresponding authors from Scopus January 1, 2017 and march 20, 2020:
  All ("surgery") AND subj ("medi") and key ("transplantation"), All ("critical care") AND subj ("medi") and key ("transplantation"), All ("ethics") AND subj ("medi") and key ("transplantation"). B. Emailing through the mailing list of scientific societies. C. The link to the survey published online. D. The link to the survey circulated through personal contacts and via social media sites.

SUMMARY:
Background COVID-19 has brought into questioning the equitable distribution of resources. Solid Organ Transplants (SOT) are life-saving procedures. Rapid changes in the management of patients are occurring, with potential for inequity. Drawing on professionals across transplant specialities, we investigated resource distribution specifically for SOT to guide healthcare policies.

A multidisciplinary team developed a survey. The survey included demographic questions to contextualise respondents, questions on resource allocation for SOT. Multiple strategies were used to distribute the survey internationally. Descriptive, uni-multivariate ordinal regressions analysis were performed. Open comments were analysed using qualitative methods.

ELIGIBILITY:
Inclusion Criteria:

* transplant surgeons, referring doctors, transplant physicians, transplant coordinators, transplant ICU doctors, COVID-19 ICU, Infectious Disease Doctors, Pulmonologists, Internist, and Ethicists

Exclusion Criteria:

* not applicable

Age Groups: Child, Adult, Older Adult
Study Population: Country macro regions, subspecilaties and organ of interest
Sampling Method: Non-Probability Sample
Enrollment: 1819 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Management of Solid Organ Transplant during COVID-19 pandemic | 20/04/2020
  Question 1"Given the COVID-19 outbreak, should liver transplant activities be stopped?" with three possible answers (Completely, Selectively and Not at All)
Equity of resource distribution | 20/04/2020
  Question 2"I feel that the current policy to allocate most resources to COVID-19 meets the equity of access in healthcare for different diseases" with four possible alternative answers (strongly agree, partially agree, partially disagree and strongly disagree).

SECONDARY OUTCOMES:
Equity rank of resource distribution | 20/04/2020
  Scale (10 strongly agree- 0 strongly disagree).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "Agostino Gemelli", Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ritschl PV, Nevermann N, Wiering L, Wu HH, Moroder P, Brandl A, Hillebrandt K, Tacke F, Friedersdorff F, Schlomm T, Schoning W, Ollinger R, Schmelzle M, Pratschke J. Solid organ transplantation programs facing lack of empiric evidence in the COVID-19 pandemic: A By-proxy Society Recommendation Consensus approach. Am J Transplant. 2020 Jul;20(7):1826-1836. doi: 10.1111/ajt.15933. Epub 2020 May 10. PMID 32323460
- [Result] The Lancet. India under COVID-19 lockdown. Lancet. 2020 Apr 25;395(10233):1315. doi: 10.1016/S0140-6736(20)30938-7. No abstract available. PMID 32334687
- [Result] Redelmeier DA, Shafir E. Pitfalls of judgment during the COVID-19 pandemic. Lancet Public Health. 2020 Jun;5(6):e306-e308. doi: 10.1016/S2468-2667(20)30096-7. Epub 2020 Apr 23. No abstract available. PMID 32334647
- [Result] Leon DA, Shkolnikov VM, Smeeth L, Magnus P, Pechholdova M, Jarvis CI. COVID-19: a need for real-time monitoring of weekly excess deaths. Lancet. 2020 May 2;395(10234):e81. doi: 10.1016/S0140-6736(20)30933-8. Epub 2020 Apr 22. No abstract available. PMID 32333839